CLINICAL TRIAL: NCT02879812
Title: Allocation System for Changes in Equity in kidNey Transplantation (ASCENT) Study
Brief Title: Disparities in National Kidney Allocation Policy
Acronym: ASCENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Rachel Patzer, Adjunct Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00081580; 1R01MD010290-01 (NIH)
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Kidney Disorders
Keywords: Transplantation Surgery; Nephrology; Organ and Tissue Transplantation; End stage renal disease (ESRD)
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Component Intervention (Experimental): End Stage Renal Disease (ESRD) facilities will receive feedback reports containing facility specific data, an educational webinar for dialysis facility medical directors and staff, and an educational video for patients and staff.
  Interventions: Other: Performance Feedback Reports; Other: Educational Video for Staff; Other: Educational Video for Patients; Other: Educational Webinar; Other: United Network for Organ Sharing (UNOS) Pamphlet
- Standard Care + Pamphlet (Active Comparator): End Stage Renal Disease (ESRD) facilities will conduct usual care and receive United Network for Organ Sharing (UNOS) educational pamphlets for staff.
  Interventions: Other: Standard Care; Other: United Network for Organ Sharing (UNOS) Pamphlet

INTERVENTIONS:
Other: Performance Feedback Reports — Medical directors will be provided performance feedback reports that are a summary of clinical performance of transplant and racial disparity performance over a period of time aimed at providing information to allow them to assess and adjust their transplant performance. The report will emphasize tailored facility-specific information on the mean time on dialysis for patients in that facility and transplant access performance measures, such as wait listing and transplantation, including the magnitude of racial disparity, detailing when a facility is performing below the national or regional average.
  Other Names: Audit and Feedback Report
  Arms: Multi-Component Intervention
Other: Educational Video for Staff — Dialysis facility staff will watch a ~10 minute educational video that describes the role of dialysis staff in improving transplant access, the new kidney allocation policy, and how the new policy impacts minority patients and those on dialysis for a substantial period of time.
  Arms: Multi-Component Intervention
Other: Educational Video for Patients — Dialysis facilities will receive a ~10 minute educational video targeted to dialysis patients to explain the transplant process and allocation policy.
  Arms: Multi-Component Intervention
Other: Educational Webinar — Education for medical directors and facility staff about the kidney allocation policy will be discussed in a webinar and information will be hosted on a website for participants to access. The seminar will be roughly 45 minutes, and continuing medical education (CME) credits will be offered.
  Arms: Multi-Component Intervention
Other: Standard Care — Dialysis facilities will conduct standard or usual care and education regarding transplantation.
  Arms: Standard Care + Pamphlet
Other: United Network for Organ Sharing (UNOS) Pamphlet — Dialysis facility staff will be provided an educational pamphlet detailing the changes in the new kidney allocation policy .

SUMMARY:
The purpose of the current study is to test a systems-level approach to disseminate a multicomponent, multilevel intervention consisting of educational materials about transplantation and the new kidney allocation system targeting dialysis facility medical directors, staff, and patients. Roughly 750 dialysis facilities in up to 18 End Stage Renal Disease Network regions across the United States will be randomized to receive intervention materials. The overall goal of the study is to extend the influence of the national allocation policy in reducing disparities in early steps in kidney transplant access.

DETAILED DESCRIPTION:
The purpose of the Allocation System for Changes in Equity in kidNey Transplantation (ASCENT) study is to test a systems-level approach to disseminate a multi-component intervention consisting of in the era of the new national kidney allocation policy and educational materials targeting dialysis facility medical directors, staff, and patients. The investigators will randomize ~750 dialysis facilities in up to 18 End Stage Renal Disease Network regions across the United States, where approximately half of facilities will receive the intervention materials and half will receive an informational brochure. This pragmatic, clinical effectiveness-implementation study will test the effectiveness of the multicomponent, multilevel interventions consisting of a tailored, facility-specific transplant and disparity performance report, educational videos for staff and dialysis patients, and an educational webinar for dialysis facility medical directors and staff.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis facilities with at least 25 patients composed of at least 10% African American and 10% Caucasian

Exclusion Criteria:

* Dialysis facilities with wait listing rates above the national tertile

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56332 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Patzer, PhD, MPH, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urbanski M, Lee YH, Escoffery C, Buford J, Plantinga L, Pastan SO, Hamoda R, Blythe E, Patzer RE. Implementation of the ASCENT Trial to Improve Transplant Waitlisting Access. Kidney Int Rep. 2023 Nov 2;9(2):225-238. doi: 10.1016/j.ekir.2023.10.028. eCollection 2024 Feb. PMID 38344743
- [Background] Patzer RE, Smith K, Basu M, Gander J, Mohan S, Escoffery C, Plantinga L, Melanson T, Kalloo S, Green G, Berlin A, Renville G, Browne T, Turgeon N, Caponi S, Zhang R, Pastan S. The ASCENT (Allocation System Changes for Equity in Kidney Transplantation) Study: a Randomized Effectiveness-Implementation Study to Improve Kidney Transplant Waitlisting and Reduce Racial Disparity. Kidney Int Rep. 2017 May;2(3):433-441. doi: 10.1016/j.ekir.2017.02.002. Epub 2017 Feb 9. PMID 28845470
- [Result] Patzer RE, Zhang R, Buford J, McPherson L, Lee YH, Urbanski M, Li D, Wilk A, Paul S, Plantinga L, Escoffery C, Pastan SO. The ASCENT Intervention to Improve Access and Reduce Racial Inequalities in Kidney Waitlisting: A Randomized, Effectiveness-Implementation Trial. Clin J Am Soc Nephrol. 2023 Mar 1;18(3):374-382. doi: 10.2215/CJN.0000000000000071. Epub 2023 Feb 8. PMID 36764664
- [Result] Magua W, Basu M, Pastan SO, Kim JJ, Smith K, Gander J, Mohan S, Escoffery C, Plantinga LC, Melanson T, Garber MD, Patzer RE. Effect of the ASCENT Intervention to Increase Knowledge of Kidney Allocation Policy Changes Among Dialysis Providers. Kidney Int Rep. 2020 Jul 2;5(9):1422-1431. doi: 10.1016/j.ekir.2020.06.027. eCollection 2020 Sep. PMID 32954067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of dialysis facilities began in September 2016. Data collection via surveillance data from patients of the dialysis facilities occurred retroactively for both study periods. The baseline period includes patients seen at dialysis facilities during January 2016 to December 2016, while the follow-up period includes patients seen at dialysis facilities during April 2017 to March 2018. Data collection from surveillance data concluded on August 2, 2019.
Pre-assignment Details: Information on patients seen during the study periods was obtained via surveillance data from study dialysis facilities. Only minimal information was collected about dialysis facility patients, thus, the total number of discrete patients is unknown as individuals could have been a patient of a dialysis facility during both study periods.
Units Other Than Participants: Facilities
Groups:
- Allocation System Changes for Equity in Kidney Transplantation (ASCENT) Intervention: ASCENT is a multi-component educational intervention delivered to dialysis facilities. End Stage Renal Disease (ESRD) facilities received performance feedback reports containing facility specific data, an educational webinar for dialysis facility medical directors and staff, an educational video for patients and staff; and the United Network for Organ Sharing (UNOS) pamphlet for dialysis facility staff detailing the changes in the new kidney allocation policy. The study intervention period occurred January 2017 through March 2017.
- Standard Care Plus Educational Pamphlet: Dialysis facilities randomized to the control study arm delivered standard or usual care and education regarding transplantation. Dialysis facility staff were provided the United Network for Organ Sharing (UNOS) educational pamphlet detailing the changes in the new kidney allocation policy. The study intervention period occurred January 2017 through March 2017.
Period: Baseline/Pre-intervention Period
Arm/Group | Allocation System Changes for Equity in Kidney Transplantation (ASCENT) Intervention | Standard Care Plus Educational Pamphlet
Started (Dialysis facilities randomized to a study intervention and current patients of those facilities. Data for the baseline/pre-intervention period were collected from surveillance data for patients of the dialysis facilities during January to December 2016.) | 28246; 329 Facilities (319 facilities are included in the intention to treat analyses.) | 28086; 320 Facilities (313 facilities are included in the intention to treat analyses.)
Completed | 28246; 329 Facilities | 28086; 320 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities
Period: Post-intervention Follow-up Period
Arm/Group | Allocation System Changes for Equity in Kidney Transplantation (ASCENT) Intervention | Standard Care Plus Educational Pamphlet
Started (Dialysis facilities remaining in the study and the and the patients receiving care at those facilities at the time the follow-up assessments. Data for the post-intervention follow-up study period were collected from surveillance data for patients of the dialysis facilities during April 2017 to March 2018.) | 28270; 327 Facilities (318 facilities are included in the intention to treat analyses.) | 28216; 319 Facilities (311 facilities are included in the intention to treat analyses.)
Completed | 28270; 327 Facilities | 28216; 319 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes demographics for patients of the study dialysis centers during the baseline/pre-intervention time period.
Units Other Than Participants: Facilities
Groups:
- ASCENT Intervention: ASCENT is a multi-component educational intervention delivered to dialysis facilities. End Stage Renal Disease (ESRD) facilities received performance feedback reports containing facility specific data, an educational webinar for dialysis facility medical directors and staff, an educational video for patients and staff; and the United Network for Organ Sharing (UNOS) pamphlet for dialysis facility staff detailing the changes in the new kidney allocation policy. The study intervention period occurred January 2017 through March 2017.
- Total: Total of all reporting groups
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet | Total
Number analyzed (Participants) | 28246 | 28086 | 56332
Number analyzed (Facilities) | 329 | 320 | 649
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (15.6) | 59.2 (15.6) | 59.3 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12432 | 12689 | 25121
  Male | 15814 | 15397 | 31211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4270 | 3371 | 7641
  Not Hispanic or Latino | 23976 | 24715 | 48691
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 145 | 93 | 238
  Asian | 725 | 489 | 1214
  Native Hawaiian or Other Pacific Islander | 226 | 176 | 402
  Black or African American | 10821 | 12092 | 22913
  White | 16270 | 15178 | 31448
  More than one race | 59 | 58 | 117
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28246 | 28086 | 56332

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Incident Patients Waitlisted
Description: The adjusted mean proportions of incident (new) patients waitlisted for kidney transplantation at study dialysis facilities, at the baseline and post-intervention time periods, were calculated. Incident patients are those who initiated dialysis treatment at study facilities during one of the study time periods. Mean proportions were adjusted for time and facility-level random effects.
Time Frame: Baseline (the twelve month period prior to the intervention), Post-intervention (the twelve month period after the intervention)
Population: This analysis included incident patients among the facilities included in the intention-to-treat analysis. Incident patients participated in either the baseline or post-intervention assessment. The overall number of participants analyzed is the sum of incident patients in facilities randomized to each study arm at the baseline and post-intervention periods.
Measure: Mean (95% Confidence Interval); unit: adjusted mean proportion of patients
Units Other Than Participants: Facilities
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
Number analyzed (Participants) | 11557 | 12066
Number analyzed (Facilities) | 319 | 313
adjusted mean proportion of patients
  Patients on the waitlist during the baseline time period: number analyzed (Participants) | 5915 | 6170
  Patients on the waitlist during the baseline time period | 1.39 [1.33 to 1.45] | 1.33 [1.27 to 1.39]
  Patients on the waitlist during the post-intervention time period: number analyzed (Participants) | 5642 | 5896
  Patients on the waitlist during the post-intervention time period: number analyzed (Facilities) | 318 | 311
  Patients on the waitlist during the post-intervention time period | 1.25 [1.19 to 1.31] | 1.30 [1.24 to 1.35]

2. Primary Outcome: Proportion of Black and White Incident Patients Waitlisted
Description: The adjusted mean proportions of Black versus White incident patients waitlisted for kidney transplantation at study dialysis facilities, at the baseline and post-intervention follow-up assessments, were calculated. Mean proportions were adjusted for time and facility-level random effects.
Time Frame: as for outcome 1
Population: This analysis included incident patients among the facilities included in the intention-to-treat analysis. Incident patients participated in either the baseline or post-intervention time periods. The overall number of participants analyzed is the sum of incident patients in facilities randomized to each study arm at the baseline and post-intervention assessment periods.
Measure: Mean (95% Confidence Interval); unit: adjusted mean proportion of patients
Units Other Than Participants: Facilities
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
Number analyzed (Participants) | 54213 | 54638
Number analyzed (Facilities) | 319 | 313
adjusted mean proportion of patients
  Black patients on the waitlist the the baseline time period: number analyzed (Participants) | 10821 | 12092
  Black patients on the waitlist the the baseline time period | 0.87 [0.82 to 0.93] | 1.12 [1.06 to 1.17]
  Black patients on the waitlist during the post-intervention time period: number analyzed (Participants) | 10681 | 11928
  Black patients on the waitlist during the post-intervention time period: number analyzed (Facilities) | 318 | 311
  Black patients on the waitlist during the post-intervention time period | 1.07 [1.02 to 1.13] | 1.15 [1.09 to 1.20]
  White patients on the waitlist during the baseline time period: number analyzed (Participants) | 16270 | 15178
  White patients on the waitlist during the baseline time period | 1.54 [1.48 to 1.59] | 1.42 [1.36 to 1.47]
  White patients on the waitlist during the post-intervention time period: number analyzed (Participants) | 16441 | 15440
  White patients on the waitlist during the post-intervention time period: number analyzed (Facilities) | 318 | 311
  White patients on the waitlist during the post-intervention time period | 1.27 [1.22 to 1.33] | 1.37 [1.32 to 1.42]

3. Primary Outcome: Proportion of Prevalent Patients Waitlisted During the Baseline Period
Description: The adjusted mean proportions of prevalent patients waitlisted for kidney transplantation at study dialysis facilities during the baseline time period were calculated. Mean proportions were adjusted for time and facility-level random effects.
Time Frame: Baseline (the twelve month period prior to the intervention)
Population: This analysis includes patients of the study facilities during the baseline (pre-intervention) time period.
Measure: Mean (95% Confidence Interval); unit: adjusted mean proportion of patients
Units Other Than Participants: Facilities
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
Number analyzed (Participants) | 28246 | 28086
Number analyzed (Facilities) | 329 | 320
adjusted mean proportion of patients | 2.68 [2.59 to 2.77] | 2.72 [2.63 to 2.81]

4. Primary Outcome: Proportion of Prevalent Patients Waitlisted During the Post-Intervention Time Period
Description: The adjusted mean proportions of prevalent patients waitlisted for kidney transplantation at study dialysis facilities during the post-intervention period were calculated. Mean proportions were adjusted for time and facility-level random effects.
Time Frame: Post-intervention (the twelve month period after the intervention)
Population: This analysis includes patients of study facilities during the post-intervention time period.
Measure: Mean (95% Confidence Interval); unit: adjusted mean proportion of patients
Units Other Than Participants: Facilities
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
Number analyzed (Participants) | 28270 | 28216
Number analyzed (Facilities) | 327 | 319
adjusted mean proportion of patients | 2.75 [2.66 to 2.84] | 2.56 [2.47 to 2.65]

5. Primary Outcome: Proportion of Black and White Prevalent Patients Waitlisted During the Baseline Period
Description: Waitlisting disparity is assessed as the adjusted mean proportion of Black versus White prevalent patients waitlisted for kidney transplantation at study dialysis facilities during the baseline time period. Mean proportions were adjusted for time and facility-level random effects.
Time Frame: Baseline (the twelve month period prior to the intervention)
Population: This analysis includes Black and White patients of study facilities during the baseline (pre-intervention) time period.
Measure: Mean (95% Confidence Interval); unit: adjusted mean percentage of patients
Units Other Than Participants: Facilities
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
Number analyzed (Participants) | 27091 | 27270
Number analyzed (Facilities) | 329 | 320
adjusted mean percentage of patients
  Black patients on the waitlist during the baseline time period: number analyzed (Participants) | 10821 | 12092
  Black patients on the waitlist during the baseline time period | 2.52 [2.43 to 2.61] | 2.71 [2.62 to 2.80]
  White patients on the waitlist during the baseline time period: number analyzed (Participants) | 16270 | 15178
  White patients on the waitlist during the baseline time period | 2.66 [2.57 to 2.75] | 2.67 [2.58 to 2.76]

6. Secondary Outcome: Knowledge About the Kidney Allocation System
Description: Knowledge about the kidney allocation system was assessed using a survey among dialysis facility medical directors or nurse managers. The survey measured provider knowledge of Kidney Allocation System (KAS) and transplantation using a cumulative knowledge score ranging from 0 to 5, where 0 = least knowledge and 5 = highest level of knowledge (higher scores are preferable, indicating greater knowledge).
Time Frame: Baseline, Immediately Post-intervention (3 months after the start of the intervention)
Population: This analysis includes dialysis facility staff who completed this question at the baseline and post-intervention time points. One staff member per facility completed the facility surveys at each study time point. During the course of the study some facilities were lost to follow-up and some staff members did not respond to all questions at the baseline and post-intervention assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Facilities
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
Number analyzed (Participants) | 311 | 302
Number analyzed (Facilities) | 311 | 302
score on a scale
  Baseline assessment | 2.31 (1.46) | 2.45 (1.43)
  Post-intervention assessment | 3.41 (1.28) | 3.07 (1.24)

7. Secondary Outcome: Percentage of Facilities With Increases or No Change/Decreases in Staff Training
Description: Staff training about kidney transplant and the allocation system was assessed among dialysis facility medical directors or nurse managers by asking "what proportion of staff have you trained regarding the new kidney allocations system?" The staff training score was based on facility-level average percent and used a scale of 0 = 0% of staff trained, 1 = 1-20% of staff trained, 2 = 21-40% of staff trained, 3 = 41-60% of staff trained, 4 = 61-80% of staff trained, and 5 = 81-100% of staff trained. Facilities were grouped as either having an increase in the percentage of staff who were trained about KAS, or had no change or a decrease in the percentage of staff trained between the baseline and post-intervention follow-up at 3 months.
Time Frame: Baseline, Immediately Post-intervention (3 months after the start of the intervention)
Population: as for outcome 6
Measure: Number; unit: Percentage of facilities
Units Other Than Participants: Facilities
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
Number analyzed (Participants) | 259 | 251
Number analyzed (Facilities) | 259 | 251
Percentage of facilities
  Facilities with increases in staff training from baseline to post-intervention | 76 | 72
  Facilities with no change or a decrease in staff training from baseline to post-intervention | 24 | 28

8. Secondary Outcome: Percentage of Facilities With Increases or No Change/Decreases in Patient Education
Description: Patient education about kidney transplant and the allocation system was assessed among dialysis facility medical directors or nurse managers by asking "what proportion of patients in this specific facility have you or your staff educated about kidney transplantation?" The patient education score was based on facility-level average percent and recorded as ordinal responses scored on a scale of 0 = 0% of patients educated, 1 = 1-20% of patients educated, 2 = 21-40% of patients educated, 3 = 41-60% of patients educated, 4 = 61-80% of patients educated, and 5 = 81-100% of patients educated. Facilities were grouped as either having an increase in the percentage of patients educated about KAS, or had no change or a decrease in the percentage of patients educated between the baseline and post-intervention follow-up at 3 months.
Time Frame: Baseline, Immediately Post-intervention (3 months after the start of the intervention)
Population: as for outcome 6
Measure: Number; unit: Percentage of facilities
Units Other Than Participants: Facilities
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
Number analyzed (Participants) | 288 | 281
Number analyzed (Facilities) | 288 | 281
Percentage of facilities
  Facilities with increases in patient education from baseline to post-intervention | 46 | 54
  Facilities with no change or a decrease in patient education from baseline to post-intervention | 54 | 46

9. Secondary Outcome: Percentage of Facilities With Increases or No Change/Decreases in Intent to Refer Patients for Kidney Transplantation
Description: Change in referral practices were measured by asking dialysis facility medical directors or nurse managers about the estimated number of patients where were referred for kidney transplantation in that facility. The medical director or nurse manager was asked "since the beginning of the ASCENT quality improvement project (about 3 months ago), have you been referring more or fewer patients?" Possible responses were: more, same, fewer, or unsure. Facilities were grouped as either having an increase in the number of patients referred for transplant, or had no change or a decrease in the proportion of patients referred for transplant.
Time Frame: Immediately Post-intervention (3 months after the start of the intervention)
Population: as for outcome 6
Measure: Number; unit: Percentage of facilities
Units Other Than Participants: Facilities
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
Number analyzed (Participants) | 295 | 292
Number analyzed (Facilities) | 295 | 292
Percentage of facilities
  Facilities with increased intent to refer for transplant from baseline to post-intervention | 27 | 23
  Facilities with same or decreased intent to refer for transplant from baseline to post-intervention | 73 | 77

10. Primary Outcome: Proportion of Black and White Prevalent Patients Waitlisted During the Post-Intervention Time Period
Description: Waitlisting disparity is assessed as the adjusted mean proportion of Black versus White prevalent patients waitlisted for kidney transplantation at study dialysis facilities during the post-intervention period. Mean proportions were adjusted for time and facility-level random effects.
Time Frame: Post-intervention (the twelve month period after the intervention)
Population: This analysis includes Black and White patients of study facilities during the post-intervention time period.
Measure: Mean (95% Confidence Interval); unit: adjusted mean percentage of patients
Units Other Than Participants: Facilities
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
Number analyzed (Participants) | 27122 | 27368
Number analyzed (Facilities) | 327 | 319
adjusted mean percentage of patients
  Black patients on the waitlist during the post-intervention time period: number analyzed (Participants) | 10681 | 11928
  Black patients on the waitlist during the post-intervention time period | 2.78 [2.69 to 2.87] | 2.56 [2.47 to 2.65]
  White patients on the waitlist during the post-intervention time period: number analyzed (Participants) | 16441 | 15440
  White patients on the waitlist during the post-intervention time period | 2.69 [2.60 to 2.78] | 2.51 [2.42 to 2.60]

ADVERSE EVENTS:
Time Frame: Information about adverse events was not collected during this study.
Description: Health information was not collected from patients receiving dialysis at the study dialysis centers at any time during the study.
Arm/Group | ASCENT Intervention | Standard Care Plus Educational Pamphlet
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT02879812/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT02879812/ICF_001.pdf